CLINICAL TRIAL: NCT01748136
Title: Screening for Lung Cancer in the HIV Patient
Acronym: NA_00036809
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Other Study IDs: J0491; NA_00036809 (Other: JHMIRB)
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Lung Cancer in the HIV Patient; HIV Infections; HIV Seropositivity; Lung Cancer
MeSH Terms: conditions — HIV Infections; HIV Seropositivity; Lung Neoplasms | interventions — Tomography, X-Ray Computed; Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single Arm: CT Scan Arm
  Interventions: Device: CT Scan with Spirometry

INTERVENTIONS:
Device: CT Scan with Spirometry — During the screening and later during the five annual study visits the patients will be scheduled to undergo total of five CT scans. The first CT scan will take place at the beginning of the study and then each year for a period of five years.

SUMMARY:
That computed tomography (CT) screening of HIV-seropositive heavy smokers will detect early stage lung cancer at significantly higher rates than what is currently being observed.

DETAILED DESCRIPTION:
The study design is that of a prospective cohort study in which 200 smoking participants will be recruited from an existing HIV-seropositive cohort of 800 patients (the Human Oral Papillomavirus Etiology (HOPE) Study). Participants will be enrolled from the Johns Hopkins HIV (Moore) Clinic and the resources of the Johns Hopkins Adult Outpatient General Clinical Research Center (GCRC) and pilot project funding from the Lung Cancer SPORE will be utilized to fund the costs of the CT scans. An interdisciplinary team with expertise in HIV-associated malignancy, CT screening, lung cancer surgery, HIV infection, epidemiology and biostatistics has been assembled to test the hypothesis by accomplishing the following Specific Aims:

ELIGIBILITY:
* Age over 25 years old.
* Confirmed HIV seropositive by ELISA assay
* No woman who has a positive serum pregnancy
* Current or previous cumulative cigarette smoking history of > 20 pack years
* Former smokers must have quit smoking within the previous 15 years.
* No medical or psychiatric condition precluding informed medical consent.
* Ability to lie on the back with arms raised over the head.
* No metallic implants or metallic devices in the chest or back (pacemakers or Harrington rods, etc.) that would cause sufficient beam hardening artifact.
* No prior history of lung cancer.
* No prior removal of any portion of the lung, excluding percutaneous lung biopsy.
* No requirement for home oxygen supplementation for respiratory conditions.
* No participation in cancer prevention trials except smoking cessation programs
* No pneumonia or acute respiratory infection within 12 weeks of enrollment that was treated with antibiotics under physician supervision.
* No individuals within 6 months of receipt of cytotoxic agents for any condition.
* No chest CT scan within the preceding 6 months
* Signed study-specific informed consent prior to study entry.

Ages: 26 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-positive participants enrolled from the Johns Hopkins HIV (Moore) Clinic, as well as from the existing HIV-seropositive cohort of 800 patients (the Human Oral Papillomavirus Etiology (HOPE) Study).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2006-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Stage distribution of HIV-seropositive patients | Day 1
  To determine differences in stage distribution of HIV-seropositive patients at lung cancer diagnosis between those who are screened by spiral CT and historic controls.

SECONDARY OUTCOMES:
To create a specimen bank of serum, sputum, and tissue | 5 years
  To create a specimen bank of serum, sputum, and tissue from the cohort of heavy smokers with HIV at high risk for lung cancer identified in Specific Aim 1.

OTHER OUTCOMES:
Epigenetic analysis of sera and sputa | 4 weeks
  To use epigenetic analysis of sera and sputa collected in Specific Aim 2 from patients screened in Specific Aim 1 as a complementary approach to low dose helical CT in order to discriminate radiologically indeterminate nodules as either molecularly positive or negative.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Brock, MD, Principal Investigator — Johns Hopkins University